CLINICAL TRIAL: NCT02625714
Title: A Randomized, Open-label, Oral Multiple Dosing, Two-way Crossover Clinical Trial to Evaluate the Safety/Tolerability and Pharmacokinetic Profiles of SID142 in Healthy Volunteers
Brief Title: Safety/Tolerability and Pharmacokinetic Study of SID142
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SK Chemicals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SID142_BE_I_2015
Record Dates: First submitted 2015-12-04; First posted 2015-12-09 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Arterial Occlusive Diseases
MeSH Terms: conditions — Arterial Occlusive Diseases | interventions — renexin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A group (Other): Renexin® → SID142
  Interventions: Drug: Renexin®; Drug: SID142
- B group (Other): SID142 → Renexin®
  Interventions: Drug: Renexin®; Drug: SID142

INTERVENTIONS:
Drug: Renexin® — Cilostazol 100mg/ginko biloba leaf extract 80mg, Immediate release, bid
Drug: SID142 — Cilostazol 200mg/ginko biloba leaf extract 160mg, Controlled release, qd

SUMMARY:
A randomized, open-label, oral multiple dosing, two-part, two-way crossover clinical trial to evaluate the safety/tolerability and pharmacokinetic profiles of SID142 in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult aged between 19 and 45
2. Weights more than 50Kg , BMI between 18.5 and 25.0 kg/m2
3. Subject without congenital or chronic disease requiring medical treatment and any pathological symptoms or opinion according to internal examination
4. Subject with acceptable laboratory result and ECG result
5. Negative result to blood serum human chorionic gonadotropin[hCG] pregnancy test at screening and urine hCG pregnancy test prior to administration in female subject. In addition, at least one condition should be corresponded which is stated below

   * Menopause(no menstruation for at least 2 years)
   * surgically sterile (hysterectomy or both oophorectomy, tubal ligation or other method)
   * Male partner should be sterile(confirmed as aspermia after deferentectomy) and sole before screening.
   * Woman who agreed to use proper method of conception accurately and continuously from at least 14 days before first Investigational Product[IP] administration to at least 30days after dosing.
6. Male subject should use contraception(condom) during clinical trial and maintain contraception and agree not to donate sperm until 28days after last dosing.
7. Subject who was given and completely understood full explanation about the study, decided to participate in the study and signed written informed consent willingly.

Exclusion Criteria:

1. Female subject who is pregnant or breast-feeding
2. Person who has anaphylaxis for IP component or clinically significant medical history of anaphylaxis for other drugs
3. Subject with a clinically significant medical history of disease on liver, kidney, nervous system, respiratory system, endocrine system, blood tumor, urinary system, cardiovascular system, musculoskeletal system or psychiatric disorder or others below

   * severe nephrotic disorder
   * moderate or severe hepatic disorder
   * menstruation period
   * aortocoronary stenosis complication
   * disease or predisposition of bleeding
   * congestive heart failure or arrhythmia
   * diabetes mellitus or glucose tolerance disorder
4. Subject with clinically significant findings on electrocardiogram[ECG] result during screening as stated below

   * QTc > 450 ms
   * PR interval > 200 msec
   * QRS duration > 120 msec
5. Active liver disease or inadequate laboratory result: AST[aspartate aminotransferase] , ALT[alanine aminotransferase] > 1.5 x upper limit of normal range
6. At screening, subject with clinically significant vital signs(sitting position blood pressure): Systolic blood pressure >140 mmHg or < 90 mmHg, diastolic pressure > 90 mmHg or < 60 mmHg
7. Hereditary galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption syndrome
8. Subject with a presence of gastroenteric disease or history of gastroenteric surgery which can influence the drug absorption
9. Subject who has been seriously injured or received surgery or shown suspicious acute disease symptoms within 4 weeks of first administration.
10. Consumption of excessive alcohol continuously or the subject who cannot quit drinking within 3 days prior to IP administration and during clinical trial period or subject who smokes
11. A history of taking any ETC drugs[Ethical drugs], oriental medicine within 2 weeks or OTC drugs[Over-the-Counter drugs] within 1week prior to first administration
12. Participation in another clinical trial in the previous 3 months before first administration of this study
13. Donation of whole blood in the previous 2 months or apheresis blood in the previous 1 month before first administration
14. The subject with abnormal diet which can influence absorption, distribution, metabolism, and excretion of drug
15. Consumption of food which can influence drug metabolism or caffeine within 48 hours after the first administration, or the subject who cannot quit consumption of such foods during whole study period.
16. Positive results to serum tests (HBsAg[hepatitis B surface antigen], anti-HCV Ab[hepatitis C virus antibody], anti-HIV Ab[human immunodeficiency virus antibody], VDRL[Venereal Disease Research Laboratory] test)

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2015-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
AUC[Area under the concentration curve]τ,ss of Cilostazol | During 144hours post-dose in each period
  Total 68 time points during periods of both 1 and 2
Cmax,ss of Cilostazol | During 144hours post-dose in each period
  Total 68 time points during periods of both 1 and 2

SECONDARY OUTCOMES:
AUClast,ss of Cilostazol | During 144hours post-dose in each period
  Total 68 time points during periods of both 1 and 2
Tmax,ss of Cilostazol | During 144hours post-dose in each period
  Total 68 time points during periods of both 1 and 2
CL[clearance]SS/F of Cilostazol | During 144hours post-dose in each period
  Total 68 time points during periods of both 1 and 2
T1/2 of Cilostazol | During 144hours post-dose in each period
  Total 68 time points during periods of both 1 and 2
Incidence rate of Adverse Events | During 25days from first administration of period 1

CONTACTS AND LOCATIONS:
Overall Officials: Min Kyu Park, MD,PhD, Principal Investigator — Dong-A University Hospital